CLINICAL TRIAL: NCT07053163
Title: Role of Low Dose of Norepinephrine Administration Within 24-Hour Mortality in Traumatic Patient With Hemorrhagic Shock
Brief Title: Low Dose of Norepinephrine Within 24-Hour Mortality in Traumatic Patient With Hemorrhagic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Radwa Gamal Said Abdeldayem, Resident, Tanta University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 36264MS298/8/24
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2023-09

CONDITIONS: Mortality Rate; Hemorrhagic Shock
Keywords: Norepinephrine; Mortality; Traumatic Patient; Hemorrhagic Shock
MeSH Terms: conditions — Shock, Hemorrhagic | interventions — Crystalloid Solutions; Blood Specimen Collection; Resuscitation; Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crystalloid and blood as resuscitation (Experimental): Patients receive crystalloid and blood as resuscitation.
  Interventions: Drug: Crystalloid and blood as resuscitation
- Crystalloid& blood and low dose of norepinephrine (Experimental): receive crystalloid, blood and low dose of norepinephrine.
  Interventions: Drug: crystalloid, blood and low dose of norepinephrine

INTERVENTIONS:
Drug: Crystalloid and blood as resuscitation — Patients receive crystalloid and blood as resuscitation
  Arms: Crystalloid and blood as resuscitation
Drug: crystalloid, blood and low dose of norepinephrine — Group 2: receive crystalloid, blood and low dose of norepinephrine
  Arms: Crystalloid& blood and low dose of norepinephrine

SUMMARY:
The aim of the work is to evaluate role of low dose of nor epinephrine administration in the early 24-hour period among traumatic patients and hemorrhagic shock. The primary outcome: evaluate mortality at first 24 hour. The secondary outcome : measure total fluid intake, observe renal functions and Hemodynamic changes.

DETAILED DESCRIPTION:
Uncontrolled hemorrhage remains the leading cause of preventable death among patients with trauma, despite considerable improvements in trauma care Trauma- induced hemorrhage and hypovolemia can trigger an increase neurohormonal response and hypotension is not explained by hypovolemia alone but is associated with sympathy inhibitory-induced vasodilation. Trauma was defined as any exposure to nonpenetrating or penetrating kinetic energy, collision, or deceleration, Patients were alive on admission with hemorrhagic shock, defined by prehospital or admission mean arterial blood pressure less than 65 mm Hg. Management of shock after trauma remains a clinical challenge, in particular if associated with active hemorrhage and vasopressors are part of the recommended therapeutic routinely used by clinicians in Europe . Historically, the importance of permissive hypotension and the restriction of crystalloid fluid volume before hemorrhage control has been confirmed with good outcomes in patients with penetrating trauma.

Vasopressors mimic the initial response to blood loss; improve venous return, coronary perfusion, and myocardial contractility. Generally, vasopressors are considered to have a negative impact on patient outcome in the management of hemorrhagic Shock, and the predominant strategy is based on permissive hypotension and low volume resuscitation.

vasopressor use in hemorrhagic Shock in humans. The use of vasopressors, such as norepinephrine for the hemodynamic management of hemorrhagic shock, may be considered in the early phase of resuscitation and is a common practice among several prehospital and hospital emergency teams in Europe. Where any surgical or interventional radiographic procedures for the immediate control of bleeding and early activation of massive transfusion protocol are always not available, the effects vasopressor administration for severe hemorrhagic shock following trauma is used to restore arterial pressure in hemorrhagic shock. Norepinephrine is a sympathomimetic agent with predominantly vasoconstrictive effects. Norepinephrine exerts both arterial and venous α-adrenergic stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 -65 Years old.
* Multiple organ injury.
* Recent trauma within 1st 24 hour.
* Mean arterial blood pressure <65 mmHg

Exclusion Criteria:

* Cardiac arrest at admission.
* Old trauma more than 24 hour.
* Severe brain or spinal injury (because of different target blood pressures).
* Death due to haemostatic failure within 6 hours of admission

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Mortality | at first 24 hour

SECONDARY OUTCOMES:
total fluid intake | at first 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Radwa Abdeldayem, Resident, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes